CLINICAL TRIAL: NCT01785030
Title: Peripheral Vasodilation in Healthy Adult Volunteers Receiving 50% Nitrous Oxide
Brief Title: Nitrous Oxide Vasodilation Healthy Adult Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Daniel S Tsze, MD, MPH, Assistant Professor of Clinical Pediatrics, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAK2807
Record Dates: First submitted 2013-02-01; First posted 2013-02-06 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Peripheral Vein Vasodilation
MeSH Terms: interventions — Nitrous Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 50% Nitrous oxide (Experimental)
  Interventions: Drug: 50% Nitrous oxide

INTERVENTIONS:
Drug: 50% Nitrous oxide

SUMMARY:
Nitrous oxide (N2O) is a gas that is normally used to take away pain and anxiety during painful medical procedures. However, one of its effects is to also make veins appear larger and more visible. This is useful when there is a patient who needs to have an intravenous (IV) needle put in their skin to give them medicine or ﬂuids, but may have veins that are very hard to see or feel. The mechanism of this observed effect is not entirely clear. The purpose of this study is to use an ultrasound to directly measure whether there is an actual change size of veins or change in blood flow in healthy adult volunteers when you give them 50% nitrous oxide, and see whether or not this change in size, or change in flow, is what causes the changes in visibility or palpability of the vein.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers.
* 19 years or older (inclusive)
* English speaking.

Exclusion Criteria:

* ASA class III or greater;
* History of, or suspected, difﬁcult airway based on physical exam, facial dysmorphism or syndrome
* Any condition in which air may be trapped in a body cavity. These include, but are not limited to:

Pneumothorax or chest injury, concurrent acute asthma exacerbation, middle ear occlusion, intestinal obstruction, ileus, or abdominal distension, sinusitis or maxillofacial injuries with potential for trapped gas, recent intraocular surgery or penetrating globe injury, air embolus, severe bullous emphysema (consider in patients with cystic ﬁbrosis), history of craniotomy in previous three weeks

* Pregnancy (1st and 2nd trimester)
* Increased intracranial pressure, impaired level of consciousness, or head injury
* Known Vitamin B12 deﬁciency
* Known MTHFR Deﬁciency (Inborn error of metabolism)
* History of bleomycin administration (note that the oxygen component of N2O administration is what interacts with bleomycin to cause pulmonary toxicity)
* Intoxication with alcohol or other drugs
* Any condition in which patient may be catecholamine-depleted (e.g. septic shock)
* Recent history of altered mental status
* Pulmonary hypertension
* Congestive heart failure.
* Trainees, including students, residents, and fellows, working in the pediatric emergency department.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Diameter of peripheral vein (mm) | 15-30 minutes at time of enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Tsze, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- NewYork Presbyterian Morgan Stanley Children's Hospital, New York, New York, United States